CLINICAL TRIAL: NCT00381329
Title: Pennsylvania Adolescent Smoking Study (PASS) - Randomized Controlled Trial Comparing Motivational Interviewing and Structured Brief Advice for the Reduction of Adolescent Cigarette Smoking
Brief Title: Pennsylvania Adolescent Smoking Study (PASStudy)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pennsylvania Department of Health (Other Government)
Collaborators: Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); Lehigh Valley Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SAP#4100027295_2
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Smoking Cessation
Keywords: Motivational Interviewing; Structured Brief Advice; Adolescent Smoking; Behavioral Intervention; Smoking; Primary Care; Tobacco
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing (MI)
- 2 (Active Comparator): Structured Brief Advice (SBA)
  Interventions: Behavioral: Structured Brief Advice (SBA)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — MI is an empirically supported, client-centered, directive method for matching counseling to an individual's readiness to change.
  Arms: 1
Behavioral: Structured Brief Advice (SBA) — SBA includes the administration of scripted, brief cessation counseling that follows standard health care smoking cessation guidelines.
  Arms: 2

SUMMARY:
The Pennsylvania Adolescent Smoking Study (PASStudy) will evaluate the effectiveness of Motivational Interviewing (MI) compared to Structured Brief Advice (SBA) to reduce cigarette smoking among adolescents who smoke. MI is a brief 5 session client-centered psychotherapeutic style intended to increase "the probability that a person will enter into, continue and adhere to a specific change strategy." This will be compared with SBA, which implements Best Practice Guidelines (i.e., 5 A's and 5 R's) and assists participants in accessing the best available resources for smoking cessation.

DETAILED DESCRIPTION:
The PASStudy is a Randomized Controlled Trial in which adolescents who smoke cigarettes will be randomized to receive either Motivational Interviewing (MI) or Structured Brief Advice (SBA). MI is an empirically supported, client-centered, directive method for matching counseling to an individual's readiness to change. Based on the principles of motivational psychology, client-centered therapy, and the Transtheoretical Model, MI represents a general and practical approach for changing behaviors by enhancing and facilitating an individual's own internally motivated change process.

SBA includes the administration of scripted, brief cessation counseling that follows standard health care smoking cessation guidelines. The counseling covers the 5As and 5Rs. The 5As are: Ask about smoking or tobacco use, Advise all smokers to stop smoking, Assess willingness to quit, Assist with cessation, and Arrange for follow-up). The 5 R's are used by clinicians to help motivate participants who are not yet ready to change to quit smoking; they are Relevance - emphasize the benefits of quitting, Risks - inform the participant of the risks of continuing in smoking, Rewards - emphasize the benefits of quitting, Road Blocks - identify barriers to cessation, and, finally, Repetition or repeating the other four R's at every encounter.

Participants in both groups will receive 5 counseling sessions over 8 weeks with the respective intervention. Participants randomized to the MI condition will receive five 45-60 minute MI sessions over the course of 8 weeks; 3 sessions occur in the office and the last 2 can be either by telephone or in the office. Participants randomized to the SBA condition will receive five 15-30 minute didactic SBA sessions over the course of 8 weeks; 3 sessions occur in the office and the last 2 can be either by telephone or in the office. Research staff will offer participants in both groups smoking reduction and cessation materials including websites, printed materials, hotlines, referrals to smoking cessation counseling programs. Participants will complete follow-up assessments at 8, 12 and 24 weeks post baseline. Self-reported smoking cessation, recorded on timeline followback calendars, will be biochemically verified via saliva cotinine tests at follow-up assessment visits. Prior to enrolling participants for randomization, each MI counselor will be certified for competence by completing the full, manualized treatment with up to 10 pilot participants.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 14 and < 19 years of age.
2. Must have smoked at least one cigarette during the past 30 days.
3. Must have smoked at least 100 cigarettes in their lifetime.
4. Fluent in English
5. Signed and dated IRB approved informed consent form (and assent form for subjects of appropriate age as required by each institution)

Exclusion Criteria:

1. Severe or profound mental retardation
2. Currently incarcerated or in a court mandated facility.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2007-09; Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of cigarettes smoked as measured by the Timeline Follow-back. | Baseline, Pre Counseling Sessions 1-5, Weeks 8, 12, 24

SECONDARY OUTCOMES:
Any reports of smoking cessation will be verified by a saliva cotinine assay. | Baseline, Counseling Sessions 1-5, Weeks 8, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Janet Audrain-McGovern, Ph.D, Study Chair — University of Pennsylvania; Deborah Moss, MD, MPH, Principal Investigator — University of Pittsburgh; Sarah Stevens, MD, MPH, Principal Investigator — Lehigh Valley Hospital; Jon Pletcher, MD, Principal Investigator — University of Pittsburgh; Pamela Murray, MD, MHP, Principal Investigator — University of Pittsburgh; Sara B Kinsman, MD, PhD, Principal Investigator — The Children's Hospital of Philadelphia/University of Pennsylvania
Locations (3):
- United States (3):
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Kalkhuis-Beam S, Stevens SL, Baumritter A, Carlson EC, Pletcher JR, Rodriguez D, Audrain-McGovern J. Participant- and study-related characteristics predicting treatment completion and study retention in an adolescent smoking cessation trial. J Adolesc Health. 2011 Oct;49(4):371-8. doi: 10.1016/j.jadohealth.2011.01.012. Epub 2011 May 24. PMID 21939867